CLINICAL TRIAL: NCT06731205
Title: Long-term Renal Prognosis of Neonatal Acute Kidney Injury: A Multicenter, Prospective Cohort Study
Brief Title: Long-term Renal Prognosis of Neonatal Acute Kidney Injury
Status: Not yet recruiting | Type: Observational
Sponsor: Guangzhou Women and Children's Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: [2024]442A01
Record Dates: First submitted 2024-12-09; First posted 2024-12-12 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Neonatal Acute Kidney Injury
Keywords: Neonatal Acute Kidney Injury; Long-Term Prognosis; Prognosis and Predictive Factors; Biomarkers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples Without DNA — Plasma and urine.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to conduct a multicenter, prospective neonatal acute kidney injury (AKI) follow-up cohort to describe the clinical characteristics of chronic kidney disease (CKD) in AKI cases within 1 year of follow-up and screen for effective biomarkers that can early warn of CKD progression. Ultimately, a neonatal AKI adverse prognosis warning model based on multidimensional data will be established to provide new data and new models for CKD management.

ELIGIBILITY:
Inclusion Criteria:

* Delivered in this hospital and subsequently admitted to the NICU during the study period;
* Diagnosed with neonatal AKI according to the 2015 KDIGO neonatal AKI criteria;
* Age <28 days.

Exclusion Criteria:

* Severe hydronephrosis diagnosed by prenatal renal ultrasound;
* Patients with congenital urinary malformations, including solitary kidney, cystic dysplasia, multicystic dysplastic kidney, renal dysplasia, and obstructive uropathy;
* Newborns who required congenital heart surgery within the first 7 days after birth;
* Newborns whose mothers had a history of renal failure;
* Death within 48 hours after birth;
* Other genetic syndromes or medical conditions were not eligible for inclusion according to the attending neonatologist's judgment.

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients who gave birth, were admitted to NICU and were diagnosed with neonatal AKI from Jan 2025 to Dec 2025 at the Women and Children's Medical Center of Guangzhou Medical University and other hospitals participating in this project.
Sampling Method: Non-Probability Sample
Enrollment: 1852 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of chronic kidney disease (CKD) | 1-3 years
  The incidence of CKD stage 3-5 (eGFR < 60 ml/min) within 1, 2, and 3 years of follow-up

SECONDARY OUTCOMES:
Mortality | 1-3 years
Incidence of renal replacement therapy | 1-3 years
Incidence of proteinuria | 1-3 years
Incidence of height retardation | 1-3 years
Incidence of hypertension | 1-3 years

IPD SHARING:
Plan to Share IPD: No